CLINICAL TRIAL: NCT01457183
Title: Bedside Pulse Lavage Irrigation Project
Brief Title: Clinical Evaluation of Bedside Pulse Lavage Irrigation Device
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Robert Galiano, Assistant Professor of Surgery, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU00037071; SP0003917 (Other Grant/Funding Number: Baxter Healthcare Corporation)
Record Dates: First submitted 2011-10-13; First posted 2011-10-21 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Healthy
Keywords: pulsed lavage; evaluate containment; evaluate tolerability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lavage group (Experimental): Healthy subjects with intact skin will be lavaged within the device in 3 locations on their bodies.
  Interventions: Device: Pulsed lavage (Stryker Pulsavac Plus)

INTERVENTIONS:
Device: Pulsed lavage (Stryker Pulsavac Plus) — Healthy subjects with intact skin will be lavaged through the device for 1 minute on 3 different sites. The stryker pulsavac plus will be used for the lavage.
  Other Names: Stryker Pulsavac Plus

SUMMARY:
This study evaluates how subjects with intact skin tolerate a water jet (psi 10-12) and how well the water stream is contained by a new containment device.

DETAILED DESCRIPTION:
Pulse lavage irrigation is an effective method of cleaning both acute and chronic wounds. The major drawback to pulse irrigation is that it is extremely messy and can easily contaminate the patient's surroundings, putting other patients and the person operating the device at risk. In order to obtain the benefits of pulse lavage, we have created a device that will contain the water spray from the lavage and protect both the patient and their surroundings. This study evaluates how well the device contains the spray from pulse lavage and how well subjects with intact skin tolerate pulse lavage when awake.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be healthy and willing to complete the study procedures.

Exclusion Criteria:

* Subjects must not have any chronic pain conditions or take any pain medications on a regular basis. Must not have any chronic wounds. Must not have any medical conditions that interfere with pain sensation. Must not have an allergy to skin adhesives. Patients must not be taking any immunosuppressive medications. Patients must not have any chronic infections.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Leak | up to 1 day
  After each lavage treatment, leak will be assessed by the presence of moisture outside of the lavage chamber. The time period of evaluation will take place immediately after the lavage. The subject will not be followed after their visit is complete.

SECONDARY OUTCOMES:
Seals | up to 1 day
  After each lavage treatment, the ability of the device to maintain appropriate seals between components will be assessed. The time period of evaluation will take place immediately after the lavage. The subject will not be followed after their visit is complete.

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Galiano, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States